CLINICAL TRIAL: NCT00776529
Title: Randomized Controlled Trial of Two Combinations of Strength and Sensorimotor Training: Effects on Strength, Power and Balance
Brief Title: Combination of Strength and Sensorimotor Training
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Applied Sciences of Western Switzerland (Other)
Responsible Party: Meng Jonas, University of Applied Sciences Western Switzerland, Valais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BA06-01
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Healthy Subjects
Keywords: sensorimotor training; Strengthening; Balance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Sensorimotor first (Experimental): In each of nine sessions: first sensorimotor exercises, then strengthening exercises
  Interventions: Other: Sensorimotor training first, followed by strength exercises
- B Sensorimotor & strength alternated (Experimental): In each of nine sessions: Strength and sensorimotor exercises alternated
  Interventions: Other: Strength exercises and sensorimotor exercises alternated

INTERVENTIONS:
Other: Sensorimotor training first, followed by strength exercises — nine sessions of one hour duration
  Arms: A Sensorimotor first
Other: Strength exercises and sensorimotor exercises alternated — nine sessions of one hour
  Arms: B Sensorimotor & strength alternated

SUMMARY:
AIM:

Strengthening and sensorimotor training (e.g with the aim to improve balance) are widely used in rehabilitation. There is little knowledge about the best ways to combine strengthening and sensorimotor training. Therefore, the investigators want to evaluate two types of combinations in healthy participants.

Interventions:

* Group A: 1.) warm-up; 2.) sensorimotor training; 3.) strength training (nine sessions in four weeks)
* Group B: 1.) warm-up; 2.) one strengthening exercise, followed by a sensorimotor exercise, alternating (nine sessions in four weeks)

Tests (Before first training and after four weeks):

* isokinetic test of knee extensors and flexors (60°/s; 120°/s; 180°/s; 240°/s.)
* squat jumps and countermovement jumps
* static balance test on an unstable underground (measured with accelerometer)
* dynamic balance: star excursion balance test, (a) on stable ground, (b) on unstable ground. Balance tests will be performed (c) in recovered state and (d) fatigue (i.e. after a fatiguing exercise).

Hypotheses

1. Group B (alternating sensorimotor and strength exercises) will improve more in the balance tests than Group A (sensorimotor first, strength afterwards).
2. Group B will improve more in the countermovement jump than Group A.
3. There will be no differences in the improvements in the strength, power and squat jump tests between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Able to perform strength and sensorimotor training
* At least 18 years old

Exclusion Criteria:

* Injury that does not allow training and testing
* Illness that does not allow training and testing
* Pregnancy
* Pain during exercising

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in Dynamic Balance measured with the Star Excursion Balance Test | From baseline to four weeks

SECONDARY OUTCOMES:
Change in height with counter-movement jump | From baseline to four weeks
Change in height with squat jump | From baseline to four weeks
Change in force development (Nm) in knee extensors and knee flexors | From baseline to four weeks
Change in Power knee extensors and knee flexors | From baseline to four weeks
Change in Static Balance (single leg stance on unstable ground) | From baseline to four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Meng, cand. BSc., Principal Investigator — University of Applied Sciences Western Switzerland Valais; Alain Amacker, cand. BSc., Principal Investigator — University of Applied Sciences of Western Switzerland
Locations (1):
- School of Physiotherapy, University of Applied Sciences Western Switzerland, Valais, Leukerbad, Valais, Switzerland